CLINICAL TRIAL: NCT04348097
Title: Comparison of Dry Needling and Activator Trigger Point Therapy on Upper Trapezius Trigger Points.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00464 Salman Sabir
Record Dates: First submitted 2020-03-06; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Activator therapy; Dry needling,; Myofascial pain; Upper trapezius.
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- activator trigger point therapy (Experimental): The Activator adjusting instrument used had force settings ranging from 1 to 6
  . For this study a force setting of 3 was used.
  Interventions: Device: Activator instrument; Device: dry needle
- Trigger point dry needling (Active Comparator): First, a tight band was held between the index finger and the thumb of the non-dominant hand and the needle (0.25-40 mm - Shen Long) was perpendicularly inserted into the muscle with the dominant hand.
  Interventions: Device: Activator instrument; Device: dry needle

INTERVENTIONS:
Device: Activator instrument — activator instrument was placed perpendicular over the identified trigger point and 10 thrusts were delivered, with a rate of one thrust per second
Device: dry needle — By wrist flexion and extension movements, the trigger point was needled in different directions and tried to elicit at least one local twitch response during the procedure and patient's familiar referral pain was tried to obtain . Each dry needling procedure lasted 1-2 minutes

SUMMARY:
The aim of this study was to compare the effects of Dry needling and Activator trigger point therapy on upper trapezius trigger points.Randomized controlled trial was conducted on Sixty-eight patients with active upper trapezius trigger points meeting the inclusion criteria i.e Age limit 20-45 both genders, presence of unilateral or bilateral upper trapezius Trigger Points. For bilateral presence of trigger points, the more painful side was selected. If more than one trigger points were present on the side to be treated, most painful trigger point was treated. Patients fulfilling essential criteria to identify the trigger points. According to Simon's criteria, which included a palpable taut band that was detected with palpation, the presence of a sensitive nodule in the taut band which was determined with algometry and referral pain. Exclusion criteria was specific neck pain, e.g. radiculopathy, systemic or inflammatory pain., evidence of spinal cord compression, recent neck surgery or trauma, long-term use of corticosteroids, anticoagulant use, e.g. Warfarin, presence of a blood coagulation disorder, contraindication for needling such as local infection, pregnancy with threatened abortion. Participants were selected by purposive sampling, group randomization using lottery method technique. All the participants were assessed using Numeric pain rating scale to measure pain, algometer to measure pain pressure threshold and inclinometer to measure cervical lateral flexion range of motion. A demographic form was used to collect data from patients. Patients were randomly assigned in dry needling and activator therapy group. Treatment was given at a frequency of 2 sessions per week and total 6 sessions were given to both group during a course of 3 weeks. The data was analyzed using SPSS 21.

DETAILED DESCRIPTION:
A myofascial trigger point (TrP) has been described as a hyperirritable spot located in a taut band of muscle; or a small pea or rope-like nodular or crepitant (crackling, grating) area within the muscle, which is painful to palpation or compression and refers pain, tenderness, or an autonomic response to a remote area. Some investigators stated that when pressure is applied to a TrP, a -jump sign‖ or -jump response‖ is elicited whereby the patient reacts with facial grimacing or by jumping away from the examiner.Patients with myofascial trigger points are generally characterized by the presence of one or more of the following symptoms: local pain, referred pain according to a typical pattern, pain when exerting compression or stretch on the muscle, local twitch response (LTR) provoked by the snapping palpation of the taut band, reduced force, and decreased range of motion (ROM). A combination of these symptoms can result in less functionality and quality-of-life. As a consequence, pain, ROM, and functionality are frequently used to measure the effect of treatment in patients with myofascial pain syndrome . Myofascial trigger points can be further differentiated as active or latent . Active and latent myofascial trigger points elicit local and referred pain, however active myofascial trigger points also reproduce patient symptoms, whereas latent myofascial trigger points do not .

Dry needling is a minimally invasive procedure in which an acupuncture needle is inserted directly into an myofascial trigger points.The advantages of dry needling are being increasingly documented and include an immediate reduction in local, referred, and widespread pain , and restoration of range of motion and muscle activation patterns.Dry needling is typically used to treat muscles, ligaments, tendons, subcutaneous fascia, scar tissue, peripheral nerves, and neurovascular bundles for the management of a variety of neuromusculoskeletal pain syndromes Chiropractic activator tool is an instrument for assisting with manipulation having cushioned head devices which require the applicator to pre - load or arm the device by pulling a handle against the action of a strong spring force.

A study was conducted in 2015 which concluded that Dry needling can be recommended to relieve myofacial trigger point pain of neck and shoulders in short and medium terms.

A study conducted in 2015 and found that There is moderate evidence that ischemic compression results in pain reduction, whereas there is strong evidence that dry needling has a positive effect on pain reduction. This decrease is greater compared with active range of motion exercises as well as no or placebo intervention A study conducted in 2014 and reported that dry needling is beneficial for decreasing pain immediately after treatment and at a 4-wk follow-up in patients with neck pain.

A research in 2019 showed that both extracorporeal shock wave therapy and dry needling can be employed to treat myofacial trigger point of the upper trapezius muscle in patients with non specific neck pain .

A research conducted in 2018 observed the changes in the ROM and neck disability index with Superficial dry needling and Deep dry needling techniques, but these changes were more significant in patients treated with Deep dry needling, especially in the follow-up periods A research in 2008 suggested that both ischaemic compression and activator trigger point therapy have an equal immediate clinically important effect on upper trapezius trigger point pain A study in 2008 suggested that activator trigger point therapy appeared to be more effective than myofascial band therapy or sham ultrasound in treating patients with non-specific neck pain and upper trapezius trigger points

ELIGIBILITY:
Inclusion Criteria:

* Age limit 20-45
* male and female .
* Presence of unilateral or bilateral upper trapezius Trigger Points.
* Patients identified with presence of trigger points.

Exclusion Criteria:

* Specific neck pain,
* Evidence of spinal cord compression
* Recent neck surgery or trauma.
* Long-term use of corticosteroids. Anticoagulant use, e.g. Warfarin. Presence of a blood coagulation disorder. Contraindication for needling such as local infection, pregnancy with threatened abortion

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | for three weeks
  The NPRS was used to measure the pain intensity of myofasial trigger points of the upper trapezius muscle . NPRS is a valid and reliable tool to assess pain. It consists of 10cm long line scale on which patient reports his/her pain from 0 (no pain) to (10 (worst possible pain)
Inclinometer | for three weeks
  PAOMPT Bubble inclinometer was used in our study. Patient was educated abot the procedure. Inclinometer was placed on patients head. Cervical lateral flexion was recorded by stabilizing the shoulder of the patient and asking him/her to bring his/her ear towards the shoulder. Reading was recorded by the tilt of fluid inside the inclinometer.
Algometer | for three weeks
  The pain pressre threshold was taken by applying vertical pressure over selected trigger point by a sixty pound baseline algometer. Pressure was increased at the rate of 1kg/cm until the patient reported the pain by saying 'yes'. 3 readings were taken at the interval of ten seconds and mean was considered as the selected measurement

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Institute of Medical Rehabilitation, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziaeifar M, Arab AM, Karimi N, Nourbakhsh MR. The effect of dry needling on pain, pressure pain threshold and disability in patients with a myofascial trigger point in the upper trapezius muscle. J Bodyw Mov Ther. 2014 Apr;18(2):298-305. doi: 10.1016/j.jbmt.2013.11.004. Epub 2013 Nov 9. PMID 24725800
- [Background] Cagnie B, Castelein B, Pollie F, Steelant L, Verhoeyen H, Cools A. Evidence for the Use of Ischemic Compression and Dry Needling in the Management of Trigger Points of the Upper Trapezius in Patients with Neck Pain: A Systematic Review. Am J Phys Med Rehabil. 2015 Jul;94(7):573-83. doi: 10.1097/PHM.0000000000000266. PMID 25768071
- [Background] Ramsey FE, Tomlanovich MC, Nowak RM. Cricothyrotomy instrumentation. JACEP. 1978 Sep;7(9):345-6. doi: 10.1016/s0361-1124(78)80362-1. No abstract available. PMID 45708
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849
- [Background] Yeganeh Lari A, Okhovatian F, Naimi Ss, Baghban AA. The effect of the combination of dry needling and MET on latent trigger point upper trapezius in females. Man Ther. 2016 Feb;21:204-9. doi: 10.1016/j.math.2015.08.004. Epub 2015 Aug 14. PMID 26304789
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642
- [Background] Jensen EV, Block GE, Ferguson DJ, DeSombre ER. Estrogen receptors in breast cancer. World J Surg. 1977 May;1(3):341-2. doi: 10.1007/BF01556853. No abstract available. PMID 883334